CLINICAL TRIAL: NCT04624594
Title: Artificial Intelligence (AI) Mobile Application Versus Health Care Provider (HCP) for Bodyweight Squats: A Randomized, Blinded, Controlled Clinical Trial
Brief Title: AI Mobile Application Versus HCP for Bodyweight Squats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Medical Fellowships (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AAAS7301
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Squat Form
Keywords: Exercise; Squat; Physical therapist; Artificial Intelligence (AI)
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence (AI) Group (Experimental): To determine baseline ability and serve as their own control, participants in both groups performed 10 bodyweight squat "control" repetitions without feedback followed by one minute of rest. Those in the AI group then performed 10 more "practice" repetitions with real-time audiovisual feedback from the app followed by one minute of rest. The AI's design provided one piece of feedback, if necessary, with a vocal statement and on-screen video per repetition (e.g. when a participant performed a squat repetition with their neck flexed downward, AI suggested keeping their head up with on-screen instruction). Participants in both groups then performed 10 "test" repetitions without feedback followed by one minute of rest.
  Interventions: Other: Artificial Intelligence Feedback
- Physical Therapist Group (Active Comparator): To determine baseline ability and serve as their own control, participants in both groups performed 10 bodyweight squat "control" repetitions without feedback followed by one minute of rest. Those in the PT group (n=15) also performed 10 "practice" repetitions with one piece of feedback per repetition, if necessary, from the PT followed by one minute of rest. Participants in both groups then performed 10 "test" repetitions without feedback followed by one minute of rest.
  Interventions: Other: Physical Therapist Feedback

INTERVENTIONS:
Other: Artificial Intelligence Feedback — AI mobile application provides feedback to participants randomized to artificial intelligence group.
  Arms: Artificial Intelligence (AI) Group
Other: Physical Therapist Feedback — PT provides feedback to participants randomized to physical therapist group.
  Arms: Physical Therapist Group

SUMMARY:
To assess if an artificial intelligence (AI) mobile application can identify and improve bodyweight squat form in adult participants when compared to a Physical Therapist (PT).

DETAILED DESCRIPTION:
Artificial intelligence (AI) is changing the way people can address their health needs. One such way related to physical exercise is AI-enabled exercise mobile application (digital coach), which uses motion tracking technology to monitor and provide real-time audio feedback on a person's exercise form. However, this AI technology has yet to be independently tested against an in-person evaluator (human coach) for its ability to improve exercise form. This study is a blinded randomized controlled trial comparing the ability of the digital coach (n=15) and a Physical Therapist (PT) human coach (n=15) to improve bodyweight squat form in 30 able-bodied volunteers age 20 - 35. Each volunteer performs 10 unassisted control squats, then 10 squats with assistive vocal feedback from either coach after each repetition, and finally 10 more unassisted test squats, all squats video-recorded. Three independent video evaluators count the number of correct squat repetitions completed by volunteers before and after intervention by the different coaches. This project is important to validate the digital coach compared to a PT human coach in a small population using a bodyweight squat for its wide applicability to daily movement patterns.

ELIGIBILITY:
Inclusion Criteria:

* Columbia University affiliate
* Aged 20 to 35 years
* Able to perform moderate bodyweight exercise for 10 minutes

Exclusion Criteria:

* Unable to provide consent

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Number of correct squats | Up to 15 minutes or completion of third set of squats
  Post-intervention improvement in squats will be determined by the number of correct squats in the third set as compared to the first set of squats.

SECONDARY OUTCOMES:
Number of squats that are identified correctly by AI | Up to 15 minutes or completion of third set of squats
  AI identification of correct and incorrect squats will be determined by the number of squats that are identified correctly by AI as compared with independent evaluators.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil K. Agrawal, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not shared with other researchers

REFERENCES:
- [Derived] Luna A, Casertano L, Timmerberg J, O'Neil M, Machowsky J, Leu CS, Lin J, Fang Z, Douglas W, Agrawal S. Artificial intelligence application versus physical therapist for squat evaluation: a randomized controlled trial. Sci Rep. 2021 Sep 13;11(1):18109. doi: 10.1038/s41598-021-97343-y. PMID 34518568